CLINICAL TRIAL: NCT01075295
Title: Prevention of Weight Gain in Early Psychoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rohan Ganguli, M.D., Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 133/2009
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Schizophreniform Disorder; Bipolar I Disorder; Bipolar II Disorder; Major Depressive Disorder; Substance-Induced Psychoses; Psychosis Not Otherwise Specified; Schizophrenia; Schizoaffective Disorder
Keywords: Schizophreniform Disorder; Schizophrenia, Schizoaffective disorder; Bipolar I Disorder; Bipolar II Disorder; Major Depressive Disorder with Psychotic Features,; Substance-Induced Psychoses; Psychosis Not Otherwise Specified; antipsychotic; weight gain; body mass index; BMI; waist circumference; WC; coronary heart disease; CHD
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Psychoses, Substance-Induced; Schizophrenia; Weight Gain; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Behavioural Intervention for the Prevention of Weight Gain
- TAU (Active Comparator)
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: Behavioural Intervention for the Prevention of Weight Gain — The intervention consists of four steps:
  * STEP 1 (Watchful Waiting): Measurement of body weight and Waist Circumference at the start (1 visit). Subjects that have a weight gain greater then or equal to 2% of their baseline weight will progress to Step 2
  * STEP 2 (Self monitoring): Self-monitoring of daily weight, daily food intake & physical activity (1 visit) Subjects that have a weight gain greater then or equal to 2% (from STEP 2) will progress to Step 3
  * STEP 3 (Nutrition & Exercise Counseling): Counseling for nutrition and physical activity (4 visits; 2 in-clinic, 2 telephone) Subjects that have a weight gain greater then or equal to 2% (from STEP 3) will progress to Step 4
  * STEP 4 (Intensive): Intensive behavioral training geared towards reducing caloric intake (4 in-clinic visits)
  Arms: Lifestyle Intervention
Other: TAU — Treatment as provided by individuals' existing healthcare providers
  Arms: TAU

SUMMARY:
The purpose of this study is to determine whether individuals with psychotic spectrum disorders ( Schizophrenia, Schizoaffective disorder,Schizophreniform Disorder, Bipolar Disorder (Type I),Bipolar Disorder (Type II),Major Depressive Disorder With Psychotic Features,Substance-Induced Psychoses,Psychosis Not-Otherwise-Specified (NOS)randomly assigned to a stepped behavioral intervention for the prevention of weight gain will experience less weight gain than individuals who receive usual care. There are several studies that have examined the effect of pharmacological and non-pharmacological behavioural approaches for weight loss in patients with psychosis, however studies examining strategies for prevention of obesity are lacking. This study is an important and novel approach to studying the problem of obesity in those with psychosis.

DETAILED DESCRIPTION:
The rates of obesity and related co-morbidities are several-fold higher in patients with psychosis than in the general population. In addition the life expectancy 20% shorter. Several lifestyle and illness-related factors have been implicated for these high rates, including weight gain associated with treatment with novel antipsychotics. The most important cause of death in psychosis patients is coronary heart disease (CHD), of which obesity is a major risk factor. As well, diabetes and its associated complications occur at high rates in persons with psychosis, and diabetes is both related to obesity and is an independent risk factor for CVD and mortality. It therefore seems reasonable to assume that prevention of obesity may lead to a reduced risk for CVD and diabetes. If the proposed intervention proves successful in preventing weight gain and reducing risk for CVD and diabetes, the quality and length of life for persons with psychosis will be vastly improved and medical costs reduced.

Specifically, we hypothesize that : 1a) a smaller proportion of those in the intervention will gain weight (2% or more) as compared to those receiving usual care, 1b) the mean weight gain of those randomized to the intervention will be less than the mean weight gain in those randomized to usual care 2) Increases in Body Mass Index (BMI) and waist circumference (WC) will be smaller in the intervention group as compared to the controls. 3) there will be smaller increases in cholesterol, triglycerides, blood glucose and insulin levels in the intervention group than in the control group. Exploratory analyses of changes in makers for systemic inflammation, and their relationship to weight, and lipid changes, will be conducted to develop novel hypotheses regarding mediators of CVD risk in psychosis.

The study will recruit sixty persons or outpatients with DSM-lV Psychosis with a BMI of < 30 kg/m², who have been treated for less than 2 years (Early SZ) and meet the other enrollment criteria. They will be randomly assigned in the allocation ratio 1:1 to either get a stepped behavioural intervention for prevention of weight gain (n=30) or treatment as usual (routine care, n=30). This will be a pragmatic clinical trial of 16-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 45 years (inclusive)
* Male or Female gender
* DSM-IV-TR diagnosis of Schizophrenia, Schizoaffective disorder,Schizophreniform Disorder, Bipolar Disorder (Type I),Bipolar Disorder (Type II), Major Depressive Disorder With Psychotic Features, Substance-Induced Psychoses, Psychosis Not-Otherwise-Specified (NOS)
* Outpatient status at the time of randomization
* Duration of antipsychotic treatment of less than 5 years
* Ability to provide informed consent
* Female patients of childbearing potential must be using a medically accepted means of contraception
* Treatment with olanzapine, clozapine, quetiapine,risperidone or paliperidone for less than 8 weeks duration at enrollment
* BMI between 18.5 and 30

Exclusion Criteria:

* Inability to give informed consent
* Currently enrolled in a weight management program
* Currently being treated with a medication to reduce weight
* Patients with unstable or active cardiovascular illnesses (myocardial infarction, congestive heart failure, etc), active or end-stage renal disease, and unstable thyroid disease, etc

Inclusion/exclusion criteria has been intentionally limited in order to maximize the generalizability of the study.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight | Measured at week 0, 4, 8 and 16
  The proportion with an increase in weight (2% or greater), from baseline to end point.

SECONDARY OUTCOMES:
Laboratory parameters | Measured at week 0 and 16
  * Fasting glucose
  * Insulin
  * Lipids

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Ganguli, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre. — http://www.camh.net/research